CLINICAL TRIAL: NCT05009589
Title: HUDDLE: Heart Health: Understanding & Diagnosing Disease by Leveraging Echocardiograms
Acronym: HUDDLE
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-07
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will screen for the presence of cardiovascular disease and provide education about the signs and symptoms of cardiovascular disease and heart disease.

ELIGIBILITY:
Key Eligibility Criteria:

1. at least 50 years of age on the day of the screening event
2. informed of the nature of the study, agrees to its provisions, and has provided written informed consent
3. does not have any conditions that would interfere with obtaining an echocardiogram of the heart

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include participants identified at pre-planned screening events for cardiovascular disease who provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Abnormal structural heart findings | 30 days
  The number of patients with abnormal structural heart findings as identified by echocardiography
Abnormal electrocardiography findings | 30 days
  The number of patients with abnormal electrocardiography findings such as rhythm disturbances, bundle branch or fascicular block, or other conduction delays
Risk factors associated with cardiovascular disease | 30 days
  Risk factors associated with cardiovascular disease including obesity (BMI and BSA calculations using height and weight) and blood pressure, along with personal and familial medical history.

CONTACTS AND LOCATIONS:
Overall Officials: E. Lee Rice, MD, Principal Investigator — Lifewellness Institute, San Diego, CA
Locations (1):
- Lifewellness Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okoh AK, Amponsah MKD, Cheffet-Walsh S, Patel M, Carfagno D, Linton D, Dimeff R, Braunreiter D, Harrington P, Brennan FH Jr, Kavinsky C, Everett M, Park B, Gunnarsson M, Snowden S, Mootz L, Koepnick T, Wheeler J, Clarke SE, Prince H, Sannino A, Grayburn P, Rice EL. Prevalence of Cardiovascular Disease and Risk Factors Among Former National Football League Players. J Am Coll Cardiol. 2024 May 14;83(19):1827-1837. doi: 10.1016/j.jacc.2024.03.371. Epub 2024 Apr 7. PMID 38593943